

**NHS Foundation Trust** 

| Charles Names and | | Use patient label Patient name: | |
|---|---|---|---|
| Sil | udy Number: | DOB: | |
| | | Hospital Number: | |
| | CONSENT FORM – parents or guardians | | |
| Titl | Title of Project: Measuring the metabolic cost of fever (IRAS Project ID 209010) | | |
| Na | Name of Researcher: Dr Samiran Ray/ Professor Mark Peters | | |
| <u>Su</u> | <u>mmary</u> | | |
| with documents of the control of the | Fever is part of the body's immune response, often triggered by infection. Fever is commonly treated with medicines such as paracetamol, mainly because people feel unwell with fever. However fever does have a role in fighting infection: it enables the rest of the immune system to function more efficiently, and may directly stop bacteria and viruses from multiplying. In most cases however treating fever does not matter because the rest of the immune system can cope well enough to fight the infection (with or without additional treatment, like antibiotics). In critically ill patients however any advantage in the fight against infection may be crucial. However in critical illness the body does have limited energy resources. In order to raise the body temperature energy is required. We do not know how much energy is required to generate a fever in critically ill children. Our study will aim to try and measure the energy required to generate a fever in a critically ill child, by measuring the levels of oxygen and carbon dioxide they breathe in and out (a method called indirect calorimetry). We do this using a machine that fits into the ventilator (breathing machine) circuit, without affecting the work of the ventilator. This will enable us to judge whether the benefits of a fever can be justified by the energy costs in the energy depleted state that is critical illness. | | |
| | | | Please initial all boxes |
| 1. | I confirm that I have read and understand the parent dated 10/10/2016 for the above study and been given the opportunity to ask questions and have had these an | a copy to keep. I have had | |
| 2. | I understand that participation is voluntary, and that I an at any time, without giving any reason and without my crights being affected. | | |

Consent form version number: 2
Consent form date of issue: 10/10/2016

[Parents/Guardians]



NILIC Foundation Trust

| Nar | ne of Person taking consent | Signature | Date/Time |
|---|---|---|---|
| | ne of Parent/Guardian/Legal<br>oresentative | Signature | <br>Date |
| | By e-mail: (address). | | |
| | By post: (address) | | |
| 6. | I would like to receive a repor | t of the study findings once th | ne research is complete: |
| 5. | I agree for my child to take pa | ırt in this research project. | |
| 4. | I consent for the non-identifial for the purpose of ethically ap | | ed with other collaborators |
| 3. | I understand that relevant se<br>collected during the study ma<br>Ormond Street Hospital NH<br>where it is relevant to my tak<br>individuals to access my child | y be looked at by responsibl<br>S Foundation Trust or fron<br>ing part in this research. I g | e individuals from Great<br>n regulatory authorities, |